CLINICAL TRIAL: NCT03908541
Title: Peripheral Inflammation and Brain Structural Alterations in Patients With Disorders of Consciousness.
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: Chronic inflammation
Record Dates: First submitted 2019-04-07; First posted 2019-04-09 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2018-08

CONDITIONS: Disorder of Consciousness
Keywords: Inflammatory markers; Magnetic resonance imaging; disorder of consciousness
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood (5 mL) was collected in a Vacutainer® tube without anticoagulant, using standardized phlebotomy procedures. Serum was prepared by centrifugation (2,000 g, 5 min, 4°C) and stored at -80°C until further analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evidence suggests that inflammatory processes are key elements in the secondary effects of severe traumatic brain injury (TBI). The present study was designed to examine whether the peripheral inflammatory markers and brain structural alterations be associated with clinical measures and primary outcome following severe TBI. We hypothesized that peripheral inflammatory markers might be correlated with voxel-based GM volumes in patients with disorder of consciousness.

DETAILED DESCRIPTION:
Background: Systemic inflammation, neurocognitive impairments, and morphologic brain changes are associated with outcome in patients with disorder of consciousness.

Objective: The aim of this study is to assess the value of peripheral inflammatory markers and brain structural alterations in the chronic phase after severe traumatic brain injury.

Methods: Serum levels of Interleukin (IL)-1β, IL-4, IL-6, IL-10, IL-13 and TNF-α were investigated in patients with chronic disorder of consciousness and healthy volunteers. Correlations were carried out between GM, WM, and CSF volumes and inflammatory cytokines levels. In addition, the Coma Recovery Scale-Revised (CRS-R) score was used to quantify the severity, and long-term recovery clinical outcome at 12 month was determined according to Glasgow Outcome Scale (GOS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 14 to 65 years old;
2. Patients had a history of sTBI;
3. Patients had awakened from a coma (indicating preserved sleep-wake cycles), including vegetative state and minimally consciousness state;
4. Patients stay unconscious for more than 1 month.

Exclusion Criteria:

1. Patients with acute infectious diseases or liver dysfunction;
2. Patients with serious diseases such as cardiac or pulmonary problems.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic disorder of consciousness were recruited at the rehabilitation units of Hangzhou Wujing Hospital (Hangzhou, Zhejiang, China).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Inflammatory cytokines | Six months
  Serum levels of Interleukin (IL)-1β, IL-4, IL-6, IL-10, IL-13 and TNF-α were investigated in patients with chronic disorder of consciousness and healthy volunteers.

SECONDARY OUTCOMES:
Gray matter volume | Six months
  The study uses voxel-based morphometry (VBM) to measure changes of gray matter volume in patients with chronic disorder of consciousness and healthy volunteers.
Coma Recovery Scale-Revised(CRS-R) | 30 minutes before blood collection
  Coma Recovery Scale-Revised (CRS-R) score was used to quantify the severity, which consists of 23 hierarchically arranged items that comprise six subscales addressing auditory, visual, motor, oromotor/verbal, communication, and arousal processes. The lowest item on each subscale represents reflexive activity, whereas the highest items represent cognitively mediated behaviors.
Glasgow Outcome Scale (GOS) | In one year
  A GOS value of <3 was considered as a bad recovery, while a GOS value of ≥3 was considered as a good recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, PhD, Principal Investigator — Department of Neurology and Brain Medical Centre The First Affiliated Hospital, School of Medicine, Zhejiang University 79 Qingchun Road, Hangzhou
Locations (1):
- Hangzhou Hospital of Zhejiang CAPR, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No